CLINICAL TRIAL: NCT07134088
Title: A Phase 1b/2 Study to Investigate the Safety, Efficacy and Pharmacokinetics of Administration of Subcutaneous (SC) Blinatumomab in Pediatric Participants With Relapsed/Refractory (R/R) and Minimal Residual Disease Positive (MRD+) B-Cell Precursor Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: A Study of Subcutaneous Blinatumomab in Children With R/R and and MRD+ B-Cell Precursor Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20220107
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory B-Cell Precursor Acute Lymphoblastic Leukemia; Minimal Residual Disease + B-Cell Acute Lymphoblastic Leukemia
Keywords: Blinatumomab; AMG 103; Relapsed/Refractory B-Cell Precursor Acute Lymphoblastic Leukemia; Minimal Residual Disease Positive B-Cell Precursor Acute Lymphoblastic Leukemia; R/R B-ALL; MRD+ B-ALL
MeSH Terms: conditions — Recurrence; Neoplasm, Residual; Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b: R/R B-ALL (Experimental): Participants with R/R B-ALL will receive blinatumomab as SC injection to determine the pediatric recommended Phase 2 dose (RP2D).
  Interventions: Drug: Blinatumomab
- Cohort Ph2-R (Experimental): Participants with R/R B-ALL will receive blinatumomab as SC injection at RP2D.
  Interventions: Drug: Blinatumomab
- Cohort Ph2-M (Experimental): Participants with MRD+ B-ALL will receive blinatumomab as SC injection at RP2D.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab will be administered as a SC injection for up to 5 cycles (each cycle will be 35 days).

SUMMARY:
The main objective of this study is to evaluate the safety and efficacy of SC blinatumomab in children below 12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥28 days to <12 years at the time of informed consent/assent.
* Lansky Performance Status (LPS) of ≥ 50%.
* For Phase 1b and Phase 2 cohort in participants with R/R B-ALL:

  * Participants with B-ALL relapsed after or refractory to any line of treatment including allogeneic hematopoietic stem cell transplant (HSCT).
  * Greater than or equal to 5% blasts in the bone marrow (BM) is considered as relapse in the BM.
* For Phase 2 cohort in participants with MRD+ B-ALL:

  * Participants with MRD+ B-ALL must have between ≥ 0.1% and < 5% blasts in the BM.
* Prior CD19-directed therapy will be allowed (with demonstrated continued CD19+ expression) if treatment ended >4 weeks prior to start of protocol therapy and no prior central nervous system (CNS) complications.
* Any Philadelphia chromosome-positive (Ph+) participant intolerant or refractory to prior tyrosine kinase inhibitors (TKIs) are eligible.

Exclusion Criteria:

* Active ALL in the CNS.
* History or presence of clinically relevant CNS pathology or event such as epilepsy, childhood seizure, paresis, aphasia, stroke, severe brain injuries, cerebellar disease, organic brain syndrome, psychosis, or severe (≥ grade 3) CNS events including immune effector cell-associated neurologic syndrome (ICANS) from prior CAR-T or other T-cell engager therapies.
* Isolated EM disease.
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement.
* Patients with Down Syndrome are not eligible for this study.
* Active acute or chronic graft versus host disease requiring systemic treatment with immunosuppressive medication.
* Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus or hepatitis C virus.
* Presence of an acute or uncontrolled chronic infection, or any other concurrent disease or medical condition that could be worsened by the treatment or interfere with the participant's ability to comply with the study protocol.
* Allogeneic HSCT within 12 weeks before the start of blinatumomab.

Ages: 28 Days to 4383 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-12-05 (Estimated); Study Completion 2030-06-18 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of Participants who Experienced Dose Limiting Toxicities (DLTs) | Up to 29 days
Phase 1b: Number of Participants who Experienced Treatment-emergent Adverse Events (TEAEs) | Up to approximately 7 months
Phase 1b: Number of Participants who Experienced Serious TEAEs | Up to 2 years and 7 months
Phase 1b: Number of Participants who Experienced Treatment-related TEAEs | Up to approximately 7 months
Phase 1b: Number of Participants who Experienced AEs of Interest (EOI) | Up to approximately 7 months
Phase 2; R Cohort: Number of Participants who had Complete Remission/Complete Remission with Partial Hematological Recovery (CR/CRh) Within the First 2 Cycles | Up to 70 days
Phase 2; M Cohort: Number of Participants who had CR with MRD Negative Response Within the First 2 Cycles | Up to 70 days
  MRD negative response = MRD level < 10^-4 (0.01%).

SECONDARY OUTCOMES:
Phase 1b: Number of Participants who had CR/CRh Within the First 2 Cycles | Up to 70 days
Phase 1b: Number of Participants who had CR Within the First 2 Cycles | Up to 70 days
Phase 1b: Number of Participants who had CR/CRh/Complete Remission with Incomplete Hematological Recovery (CRi) or Blast Free Hypoplastic or Aplastic Bone Marrow (BM) Within the First 2 Cycles | Up to 70 days
Phase 1b: Number of Participants with a MRD Negative Response Within the First 2 Cycles | Up to 70 days
  MRD negative response = MRD level < 10^-4 (0.01%).
Phase 1b: Duration of Response (DOR) | Up to 2 years and 7 months
  DOR is defined as the time from the first response of CR/CRh within the first 2 cycles until hematological relapse (Including extramedullary [EM] relapse) per investigator's assessment or death due to any cause, whichever occurs first.
Phase 1b: Maximum Concentration (Cmax) of Blinatumomab | Up to approximately 7 months
Phase 1b: Time to Maximum Concentration (Tmax) | Up to approximately 7 months
Phase 1b: Area Under the Concentration Time Curve (AUC) | Up to approximately 7 months
Phase 1b: Number of Participants with Anti-blinatumomab Antibodies | Cycle 1, Day 1 and Cycle 2, Day 1 (Cycle Duration = 35 days)
Phase 2: Number of Participants who had CR/CRh with MRD Negative Response Within the First 2 Cycles | Up to 70 days
  MRD negative response = MRD level < 10^-4 (0.01%).
Phase 2: DOR | Up to 2 years and 7 months
  DOR is defined as the time from the first response of CR/CRh within the first 2 cycles until hematological relapse (Including EM relapse) per investigator's assessment or death due to any cause, whichever occurs first.
Phase 2; R Cohort: Number of participants who had CR Within the First 2 Cycles | Up to 70 days
Phase 2; R Cohort: Number of participants who had CR/CRh/CRi and Blast Free Hypoplastic or Aplastic BM Within the First 2 Cycles | Up to 70 days
Phase 2: Overall Survival (OS) | Up to 2 years and 7 months
  OS is defined as the time from the first dose until death due to any cause.
Phase 2: Number of Participants who Experienced TEAEs, Serious TEAEs, Treatment Related TEAEs and EOIs | Up to 2 years and 7 months
Phase 2: Blinatumomab Serum Concentrations | Up to 175 days
Phase 2: Number of Participants with Anti-blinatumomab Antibodies | Cycle 1, Day 1 and Cycle 2, Day 1 (Cycle Duration = 35 days)
Phase 2; M Cohort: Number of participants who had CR/CRh/CRi and Blast Free Hypoplastic or Aplastic BM with MRD Negative Response Within the First 2 Cycles | Up to 70 days
  MRD negative response = MRD level < 10^-4 (0.01%).

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- St Jude Childrens Research Hospital, Memphis, Tennessee, United States
- Kanagawa Childrens Medical Center, Yokohami-shi, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com